CLINICAL TRIAL: NCT02533154
Title: Effect of Benzalkonium Chloride Containing Eye Drops on the Conjunctival Bacterial Flora of Dry Eye Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-280515
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAC treatment group (Experimental): 20 patients with mild or moderate dry eye syndrome receiving BAC containing Prosicca eyedrops for 1 month
  Interventions: Drug: Prosicca; Other: Bacterial culture
- non-BAC treatment group (Active Comparator): 20 patients with mild or moderate dry eye syndrome receiving preservative-free Prosicca sine eyedrops for 1 month
  Interventions: Drug: Prosicca sine; Other: Bacterial culture

INTERVENTIONS:
Drug: Prosicca — Prosicca eyedrops Dosage: on demand Route of administration: topical
  Arms: BAC treatment group
Drug: Prosicca sine — Prosicca sine eyedrops Dosage: on demand Route of administration: topical
  Arms: non-BAC treatment group
Other: Bacterial culture — bacterial cultures obtained with conjunctival swabs

SUMMARY:
Benzalkonium chloride (BAC) is a preservative, which is a component of more than 70% of topical ophthalmic drugs. Although BAC is a preservative with an excellent antibacterial spectrum, it has also been shown to induce toxic effects to the ocular surface. Several studies have indicated that BAC may also have altering effects on the bacterial flora of the conjunctiva.

Since dry eye syndrome (DES) is a very common and multifactorial disease of the ocular surface and the tear fluid resulting in tear film instability, inflammation of the ocular surface, symptoms of discomfort and visual impairment, there are many different preserved as well as preservative-free ophthalmic preparations of ocular lubricants for the treatment of DES. Unpublished data from our department shows differences between artificial tears for the treatment of DES with and without BAC in bacterial culture.

Therefore, the aim of this study is to investigate the effect of artificial tear eyedrops with and without BAC on the conjunctival bacterial flora. For this 40 patients with mild or moderate dry eye syndrome with no use of artificial tears in the 4 weeks preceding the study will be recruited and treated either with the preservative-free "Prosicca sine" eyedrops or the BAC containing "Prosicca" eyedrops for one month. Conjunctival samples will be collected of one eye of each patient before and after the 1-month treatment period to compare the conjunctival bacterial flora of the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 75 years.
* Signed and dated written informed consent.
* History of dry eye syndrome for at least 3 months
* Tear Break Up Time (BUT) ≤ 10 seconds or Schirmer I test ≤ 10 mm and ≥ 2mm
* Normal ophthalmic findings except dry eye syndrome, ametropia < 6 Dpt.
* Recommended use of topical lubricants, but no administration of topical lubricants 4 weeks preceding the first study day.

Exclusion Criteria:

* History or presence of ocular disease judged by the investigator as incompatible with the study.
* Any other topical ocular treatment than the study medication in the 4 weeks preceding the first study day and during the treatment period.
* Wearing of contact lenses.
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day.
* Participation in a clinical trial in the 3 weeks preceding the first study day.
* Pregnancy, lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07-27 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of colony forming units (CFU) in bacterial culture of conjunctival swab | 1 month

SECONDARY OUTCOMES:
Tear Break Up Time (BUT) | 1 month
Schirmer I test | 1 month
OSDI© score | 1 month
Instillation frequency | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria